CLINICAL TRIAL: NCT03554447
Title: Pentoxifylline as a New Adjuvant in Adult Patients With Major Depressive Disorder: Randomized, Double Blind, Placebo Controlled Trial.
Brief Title: Role of Pentoxifylline as an Adjuvant Therapy for Adult Patients With Major Depressive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahmoud Samy Abdallah (Other)
Responsible Party: Sponsor-Investigator, Mahmoud Samy Abdallah, Principal Investigator, Sadat City University
Organization: Sadat City University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0074/2015
Record Dates: First submitted 2018-05-31; First posted 2018-06-13 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Major Depressive Disorder
Keywords: Pentoxifylline; Anti-inflammatory; MDD; phosphodiastrase inhibitors
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Escitalopram; Tablets; Pentoxifylline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pentoxifylline group (Experimental): Escitalopram 20 mg tablet once daily for 12 week plus Pentoxifylline 400 mg tablet twice daily for 12 weeks
  Interventions: Drug: Escitalopram 20 mg tablet plus Pentoxifylline 400Mg Tablet
- Control group (Placebo Comparator): Escitalopram 20 mg tablet once daily for 12 week plus placebo tablet twice daily for 12 weeks
  Interventions: Drug: Escitalopram 20 mg tablet + Placebo

INTERVENTIONS:
Drug: Escitalopram 20 mg tablet plus Pentoxifylline 400Mg Tablet — Selective serotonin reuptake inhibitor plus phosphodiesterase inhibitor with anti-inflammatory properties
  Arms: Pentoxifylline group
Drug: Escitalopram 20 mg tablet + Placebo — Selective serotonin reuptake inhibitor plus placebo
  Arms: Control group

SUMMARY:
This study aimed to evaluate the therapeutic benefits of pentoxifylline (PTX) in treatment of adult patients with MDD as it has anti-inflammatory and phosphodiastrase inhibition activities.

DETAILED DESCRIPTION:
In this study, the investigators evaluated the potential antidepressant effect of PTX in adult patients with MDD. the investigators hypothesized that MDD patients taking add-on PTX would present greater amelioration of their depressive symptoms than patients taking add-on placebo. Furthermore, the investigators assessed the relationship between HAM-D score and several peripheral biomarkers as well as their role in diagnosis and therapeutic targets of MDD.

ELIGIBILITY:
Inclusion Criteria:

* Eighty adult outpatients with the Diagnostic and Statistical Manual of Mental Disorders-IV (DSM-IV) diagnosis of MDD based on a MINI Neuropsychiatric Interview (MINI) (American Psychiatric Association., 2000; Sheehan et al., 1998), without psychotic features and a total 17 item HAM-D score of at least 18 with item 1 (depressed mood) scored 2 or greater were eligible (Hamilton, 1960).
* Patients were requested to be free of all the psychotropic and anti-inflammatory medications for at least 4 weeks before participating in the study.

Exclusion Criteria:

* Patients with bipolar I or bipolar II disorder
* Patients with personality disorders
* Patients with eating disorders
* Patients with substance dependence or abuse
* Patients with concurrent active medical condition
* Patients with history of seizures
* Patients with history of receiving Electroconvulsive therapy (ECT)
* Patients with inflammatory disorders
* Patients with allergy or contraindications to the used medications
* Patients with finally pregnant or lactating females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-04-20 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Effect on Hamilton Depression rating scale score (HAM-D score) | 12 week
  The principal measure of the outcome was the 17-items HAM-D. Scoring is based on the 17-item scale and scores of 0-7 are considered as being normal, 8-13 suggest mild depression, 14-17 moderate depression and scores over 17 are indicative of severe depression. Remission is defined as HAM-D total score ≤ 7 (primary outcome). Treatment response is defined as ≥ 50% drop in the HAM-D total score.

SECONDARY OUTCOMES:
Effect on biological markers | 12 week
  Serum level of tumor necrosis factor alpha (TNF-α), Interleukin-6 (IL-6), Interleukin-10 (IL-10), brain derived neurotrophic factor (BDNF), 8-hydroxy-2'-deoxyguanosine (8-OHdG), and serotonin were measured at the baseline and after the treatment to evaluate the biological effects of the used medications.

CONTACTS AND LOCATIONS:
Overall Officials: Sahar El-Haggar, Ph.D, Study Director — Tanta University

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-01): https://cdn.clinicaltrials.gov/large-docs/47/NCT03554447/Prot_SAP_000.pdf